CLINICAL TRIAL: NCT07173920
Title: A Single-Center, Double-Blind, Randomized, Placebo-Controlled Clinical Study on the Efficacy and Safety of Repetitive Transcranial Magnetic Stimulation (rTMS) Under Precise Localization for Relieving Motor Symptoms of Tardive Dyskinesia
Brief Title: Single-Center, Double-Blind, Randomized, Placebo-Controlled Study on Efficacy and Safety of rTMS (With Precise Localization) in Relieving Motor Symptoms of TD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Xie Bingyan, Ms.XIE, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-08-13-4
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Tardive Dyskinesia; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Tardive Dyskinesia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treating tardive dyskinesia (TD) with active repetitive Transcranial Magnetic Stimulation (rTMS) (Experimental)
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Treating tardive dyskinesia (TD) with sham repetitive Transcranial Magnetic Stimulation (rTMS) (Placebo Comparator)
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — Patients will receive rTMS treatment for a total of 14 days. Prior to treatment, patients will undergo an MRI scan; the images will be preprocessed to construct a structural network, and precise localization of the pre-SMA (preSupplementary Motor Area) region and the SCAN (Somatosensory-Cognitive-Action Network) will be performed based on coordinates.

SUMMARY:
# Brief Summary (English Version) Tardive Dyskinesia (TD) is a hyperkinetic movement disorder induced by long-term use of dopamine receptor blockers and related drugs. Characterized by involuntary spasms or choreiform movements involving the tongue, lower face, jaw, and limbs (persisting for at least several weeks), TD causes irreversible neurological damage that persists even after discontinuing the causative drugs, significantly impairing patients' functional outcomes.

rTMS is a non-invasive neuromodulation technique: time-varying currents in a coil generate magnetic fields that penetrate the scalp and skull to act on brain neurons, inducing depolarization, neural network activation, neurotransmitter release, metabolic changes, and gene expression, thereby producing physiological effects [9]. In recent years, rTMS has gained attention for treating movement disorders (e.g., Parkinson's disease, motor neuron disease, dystonia, essential tremor, Huntington's disease) due to its non-invasiveness, high safety, and repeatability. Studies have reported that rTMS can significantly improve motor symptoms in TD patients [10, 11]; however, existing research is limited by small sample sizes, conventional treatment parameters, large inter-individual variability, and unclear long-term efficacy.

rTMS efficacy in TD is strongly influenced by parameters including stimulation targets, localization methods, sequences, and cycles. Optical navigation (using personalized MRI) is the most accurate and yields the best therapeutic effects, compared to manual localization or positioning caps . Regarding stimulation sequences, 1Hz and 20Hz rTMS have shown efficacy but with short-lived effects. Continuous theta-Burst Stimulation (cTBS)-a specialized rTMS mode that delivers rapid pulse trains mimicking endogenous theta-wave bursts-provides higher therapeutic doses in less time, enabling more durable efficacy and effectively reducing motor cortex excitability .

Therefore, this study aims to investigate the effect of cTBS (under precise localization) on improving motor symptoms in patients with TD.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age between 18 and 65 years; (2) Patients whose diagnosis is consistent with the tardive dyskinesia (TD) diagnostic criteria defined by the Schooler-Kane criteria, with a disease duration of at least 3 months before screening, and a history of treatment with dopamine receptor antagonists for at least 3 months (a minimum of 1 month for patients aged ≥ 60 years); other diseases that may cause involuntary movements are excluded

Exclusion Criteria:(1) Diagnosed with movement disorders other than tardive dyskinesia (TD); (2) A history of focal brain injury or severe leukoencephalopathy (Fazekas grade 3 or higher) identified on previous head MRI/CT; (3) A personal history of epilepsy, unexplained loss of consciousness, or current use of anticonvulsant medications for seizure management; (4) Presence of metallic medical devices in the body (e.g., cardiac pacemakers, cochlear implants), other metallic foreign bodies, or any electronic devices implanted in the body; or having other contraindications to repetitive Transcranial Magnetic Stimulation (rTMS); (5) Presence of contraindications to MRI scanning, such as having metallic implants in the body or claustrophobia

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Use the Abnormal Involuntary Movement Scale (AIMS) to assess the improvement in abnormal movements in patients with tardive dyskinesia (TD) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Sixth Hosptial, Beijing, China

IPD SHARING:
Plan to Share IPD: No